CLINICAL TRIAL: NCT02775487
Title: Smog Induced Indoor Air Pollution in Homes of Chronic Obstructive Pulmonary Disease Patients: Effectiveness of Controls
Brief Title: Smog Induced Indoor Air Pollution in Homes of Chronic Obstructive Pulmonary Disease Patients.
Status: Withdrawn | Type: Observational
Why Stopped: Withdrawn before IRB review. Investigator no longer working at facility.
Sponsor: University of Missouri-Columbia (Other)
Collaborators: University of Texas at Austin (Other)
Responsible Party: Sponsor
Other Study IDs: ST-MU-UT 2012
Record Dates: First submitted 2012-01-23; First posted 2016-05-17 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Air quality
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD and air quality: Persons enrolled in the study will have been diagnosed with Stage III or IV COPD and samples of air taken from their home environment.

SUMMARY:
Primary objective of this project is to measure the impact of passive control and active control systems on indoor pollution that is directly or indirectly related to ambient air pollution (smog). The first goal will be to measure baseline parameters for 50 homes, including information about the building, ventilation characteristics, pollution levels (indoors and outdoors), and occupant survey information. In a subset of these homes, either passive or active control systems will be installed and the impact of these systems on indoor concentrations. Participants will be enrolled on a rolling basis (5-15 persons studied at a given point in time) over a 16-month period. Participants will be followed for approximately 5 weeks and data obtained at three points in time: at enrollment (day 1 of study), after 1 week (baseline verification) and after four weeks with the control system in the home (at the end of study week 5).

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a degenerative lung disease resulting in lower lung function characterized by an obstruction to airflow. COPD is an umbrella term for two disease processes: chronic bronchitis and emphysema. It is currently the 4th leading cause of death in the United States. Approximately 14 million Americans are known to suffer from COPD; however, it is estimated that as many as 24 million Americans may have some form of one or both of the diseases (Centers for Disease Control, 2011). The primary risk factor for developing COPD is cigarette smoking; other factors include exposure to air pollution, occupational dusts and chemicals, and lower socioeconomic status. Poverty has been identified as a risk factor for COPD but the aspects related to poverty that increase the risk of COPD are unclear (GOLD, 2011). Lower education level and household income has been noted to relate to increased severity of COPD (Eisner, Blanc, Omachi, Yelin, Sidney, Katz, et al, 2011). An American Lung Association survey found that over half of those diagnosed with COPD reported that their condition limits their ability to perform activities of daily living, including activities in the home (American Lung Association, 2009). As air pollution can lead to an exacerbation of COPD symptoms and precipitate emergency room visits and hospitalization, minimizing pollution in indoor air may be a key component of disease management and decreasing health care costs.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of COPD (stage III or IV); adults over the age of 18 years

Exclusion Criteria:

* Children (persons under age 18), fetuses, neonates, pregnant women, prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited from pulmonary rehabilitation centers in St. Louis, MO. Potential participants will be screened to ascertain eligibility based on diagnosis and stage of disease progression.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in Air quality measures at week 5 | week 5 of study
  Air samples taken from the home

SECONDARY OUTCOMES:
Change in Borg scale for breathlessness from week 1 to week 5 | week 1 of study, week 2 of study and week 5 of study
  Scale on which participant rates perceived breathlessness
Change in vital signs from week 1 to week 5 | week 1 of study, week 2 of study and week 5 of study
  Heart rate, respiratory rate, blood pressure, oxygen saturation (SpO2) via pulse oximetry, bedside spirometry
Change in Air quality measures from week 1 to week 5 | week 1 and week 2 of the study
  Change in Air quality measures from week 1 to week 5

CONTACTS AND LOCATIONS:
Overall Officials: Shawna L Strickland, PhD, RRT, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No